CLINICAL TRIAL: NCT04618016
Title: Prospective, Randomized, Single-blind, Multinational, Long-term Study for the Evaluation of the Clinical Outcome, Oxidation Profile and Wear Analysis of Medium Cross-linked Polyethylene With and Without Vitamin E for Total Knee Arthroplasty
Brief Title: Evaluation of Medium Cross-linked Polyethylene With and Without Vitamin E for Total Knee Arthroplasty
Acronym: VIKEP
Status: Active, not recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Collaborators: Raylytic GmbH (Industry); B. Braun Medical France (Unknown)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1906
Record Dates: First submitted 2020-10-27; First posted 2020-11-05 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis, Knee; Arthritis, Rheumatoid; Intra-Articular Fractures; Joint Instability; Genu Valgum or Varum
Keywords: Total Knee Arthroplasty; Range of motion; Treatment outcome; Ultrahighmolecular Weight Polyethylene with Vitamin E
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis, Rheumatoid; Intra-Articular Fractures; Joint Instability; Genu Valgum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- With Vitamin E
  Interventions: Device: UHMWPE with Vitamin E
- Without Vitamin E
  Interventions: Device: UHMWPE without Vitamin E

INTERVENTIONS:
Device: UHMWPE with Vitamin E — e.motion Pro (PS and UC) with MXE gliding surface
  Groups: With Vitamin E
Device: UHMWPE without Vitamin E — e.motion Pro (PS and UC) with β-PE gliding surface
  Groups: Without Vitamin E

SUMMARY:
Prospective, randomized, single-blind, multinational, long-term study for the evaluation of the clinical outcome, oxidation profile and wear analysis of medium cross-linked Polyethylene with and without Vitamin E for total knee arthroplasty

ELIGIBILITY:
Inclusion Criteria:

* Indication for a total knee replacement with a mobile-bearing UC or PS inlay
* Written informed consent for participating at the clinical study
* Willingness and mental ability to participate at the long-term follow-up examinations

Exclusion Criteria:

* Patient age < 18 and > 80 years
* Pregnancy
* High risk patients (ASA class >3)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: multicentric
Sampling Method: Probability Sample
Enrollment: 605 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2034-10 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcome measured with the KSS [performance] | 10 years postoperatively
  The KSS is an examiner-administrated standard clinical evaluation tool reporting results for patients undergoing TKA. It separates findings in the operated knee (kKSS) score from findings related to the patient's function (fKSS), which might be affected by co-morbidities. The two sub-scores are reported separately ranging from 0 points (worst result) to 100 points (best results), as well as summarized score, total KSS. Final grading of total KSS results Scores of 160 to 200 will be rated as excellent, 140 to 159 as good, 120 to 139 as fair, and less than 120 as poor.

SECONDARY OUTCOMES:
Survival rate | until the last follow-up at 10 years postoperatively
  Kaplan-Meier Analysis is a standard statistical method to describe the survival of human subjects or medical products over a defined time period. The revision-free survival rate is the performance indicator of the product under investigation and confirms the clinical outcome of the knee prosthesis. Information on survival of the implant will be collected until the last follow-up of the study patients took place.
Progress of Clinical Outcome [Oxford Score] compared to baseline | Preoperatively, 3 months, 12 months, 3 years, 5 years, 7 years, 10 years
  The Oxford Knee Score is a reliable 12-item, patient-reported questionnaire originally developed and validated specifically to assess function and pain in patients undergoing total knee replacement. It is short, reproducible, valid and sensitive to clinically important changes over time. Each of the 12 questions on the OKS is scored in the same way with the score decreasing as the reported symptoms increase (i.e. become worse). All questions are laid out with response categories denoting least (or no) symptoms to the left of the page (scoring 4) and those representing greatest severity lying on the right hand side (scoring 0), as detailed for question 1 below. This method, when summed, produces overall scores running from 0 to 48 with 48 being the best outcome, (to convert from the 60-12 system to the 0-48 system and vice versa subtract the score from 60).
Quality of Life [EQ-5D-5L] | Preoperatively, 3 months, 12 months, 5 years, 10 years
  EQ-5D is a standardized 5-dimension 5-level measure of the health status and is developed by the EuroQol Group in order to have a simple and generic measure for clinical and economic assessment. Instructions for the user are directly included into the questionnaire and it consists of two pages. One cover five different dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression) and the other one the EQ visual Analogue Scale (EQ-VAS). The VAS scale records the self rated health status of the patient from the level "the worst health you can imagine" to "the best health you can imagine".
Comparison of Radiographic evaluation over time | baseline (assessed at discharge from hospital up to 10 days postoperatively); 3 months; 12 months; 5 years; 10 years
  Imaging will be used to evaluate the implant status as well as device condition and potential presence of device-related Adverse Events including fracture, wear, loosening or radiolucencies.
Comparison of Radiographic alignment over time | baseline (assessed at discharge from hospital up to 10 days postoperatively); 3 months; 12 months; 5 years; 10 years
  Alignment (femoral-knee baseline angle, tibial-knee baseline angle, femoral-tibial angle (mechanical))
Oxidation profile and wear analysis of available retrievals | During the course of the study up to 10 years postoperatively
  Available retrievals of explanted investigational products will be analysed by the biomechanical laboratory of the sponsor. Therefore any retrieval has to be returned to the Sponsor's facility after its revision in order to perform these analyses. Special focus of theses analyses are the oxidation profile, the wear behaviour, the mechanics and the cumulative linear abrasion of these retrievals. These measurements can further analyse the in-vivo performance of the device of the reference and investigational product
Further analysis of patients having a revision of the primary implant | During the course of the study up to 10 years postoperatively
  In case a patient requires the revision of the primary implanted knee prosthesis, additional information on the revision surgery shall be collected. The reason for revision together with the clinical symptoms shall be documented. Further examinations (e.g. arthroscopy) prior to the revision and the date of revision surgery is to be documented. If pre revision radiographs are taken as part of the clinical routine, the results of the radiographic analysis shall be documented in the respective CRF.
(Serious) Adverse Events | During the course of the study up to 10 years postoperatively
  During the course of the study, any upcoming intra- or postoperative (serious) adverse device events or effects related or not related to the product under investigation, will be documented. The total number of AEs will be summarized and further evaluated by the sponsor and reported according to local legislation and necessity. Recorded complications will be categorized and analyzed in order to assess the safety of the investigational product.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfram Mittelmeier, Prof. Dr., Principal Investigator — Orthopädische Uniklinik Rostock, Direktor
Locations (8):
- France (2):
  - Hôpital Sud - CHU de Grenoble, Échirolles, Isere
  - CHU Amiens-Picardie, Amiens
- Germany (6):
  - Lukas Krankenhaus, Bünde, North Rhine-Westphalia
  - Brüderhaus Koblenz, Koblenz, Rhineland-Palatinate
  - Park-Klinik Weißensee, Berlin
  - Waldkliniken Eisenberg, Eisenberg
  - Krankenhaus Reinbek, St. Adolf Stift, Reinbek
  - Universitätsklinikum Rostock, Klinik für Orthopädie, Rostock

REFERENCES:
- [Derived] Maier K, Selig M, Haddouche A, Haunschild M, Hauschild O, Khalili I, Kirschberg J, Lutter C, Menges M, Mertl P, Niemeier A, Rubens-Duval B, Mittelmeier W. Vitamin E-enriched medium cross-linked polyethylene in total knee arthroplasty (VIKEP): clinical outcome, oxidation profile, and wear analysis in comparison to standard polyethylene-study protocol for a randomized controlled trial. Trials. 2024 Jan 5;25(1):27. doi: 10.1186/s13063-023-07811-1. PMID 38183062